CLINICAL TRIAL: NCT06627309
Title: Rapid DFLC Response Predict Complete Hematologica Response in Systemic AL Amyloidosis Patients Treated with Daratumumab-based Regimen
Brief Title: Rapid DFLC Response Predict CHR in AL Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Principal of Investigator, Peking University People's Hospital
Other Study IDs: 2023PHB319-001-02
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Systemic AL Amyloidosis
Keywords: rapid dFLC response; daratumumab; systemic al amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Pharmaceutical Preparations; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: All patients in this cohort receive daratumumab, bortezomib and dexamethasone as treatment.
  All patients receive additional sFLC examination in C1D7, C1D14.
  Interventions: Drug: Dara IV; Drug: Bortezomib (drug); Drug: Dexamethasone; Drug: Cyclophosphamide (CTX); Drug: Dara SC

INTERVENTIONS:
Drug: Dara IV — The treament follow the clinical routine practice, as daratumumab 16mg/kg iv qw OR dara SC 1800mg initially. The treatment schedule involve weekly administrations during cycles 1 to 2, following by biweekly administrations during cycles 3 to 6. Subsequently, monthly administrations are given as monotherapy.
Drug: Bortezomib (drug) — Bortezomib is administered subcutaneously. The dosage range from 0.7 to 1.3 mg/m2 on days 1, 8, 15, and 22 of each cycle, for a maximum of 6 cycles
Drug: Dexamethasone — Dexamethasone is administered intravenously at a dose of 40 mg weekly for each cycle, for a maximum of 6 cycles. For patients over 70 years of age or with severe edema, heart failure, or uncontrolled diabetes mellitus, dexamethasone can be administered at a dose of 10-20 mg per week.
Drug: Cyclophosphamide (CTX) — Some patients may receive cyclophosphamide orally or intravenously at a dosage of 300 mg/m2 weekly.
Drug: Dara SC — The treament follow the clinical routine practice, as daratumumab 16mg/kg iv qw OR dara SC 1800mg initially. The treatment schedule involve weekly administrations during cycles 1 to 2, following by biweekly administrations during cycles 3 to 6. Subsequently, monthly administrations are given as monotherapy.

SUMMARY:
Light chain amyloidosis (AL amyloidosis) is a rare plasma cell dyscrasia characterized by the deposition of insoluble amyloid fibrils in multiple organ systems. The treatment of amyloidosis primarily relies on anti-plasma cell therapy and supportive care. The application of anti-plasma cell therapy has significantly improved outcomes in patients with AL amyloidosis. Standard first-line therapy typically includes daratumumab, bortezomib, cyclophosphamide, and dexamethasone (Dara-BCD), achieving a complete hematologic response in nearly 60% of patients.The depth and speed of the hematologic response are strongly correlated with organ response and overall survival. An early achievement of a complete hematologic response is particularly crucial in cases of AL amyloidosis characterized by significant organ involvement. The median time to a hematologic response for the daratumumab based treatment is only 7-9 days. The retrospective data showed that the hematologic response in Day 7 in Cycle 1 (C1D7) may predict the complete hematologic response rate. In order to validate the conclusion, the investigator design this prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of systemic AL amyloidosis;
2. Daratumumab, bortezomib, dexamethasone used in treatment;
3. Informed consent explained to, understood by and signed by the patient;
4. dFLC ≥ 50 mg/L;

Exclusion Criteria:

1. Fulfill with the criteria of active multiple myeloma or active lymphoplasmacytic lymphoma;
2. Presence of other tumors which is/are in advanced malignant stage and has/have systemic metastasis;
3. Severe or persistent infection that cannot be effectively controlled;
4. Presence of severe autoimmune diseases or immunodeficiency disease;
5. Patients with active hepatitis B or hepatitis C ([HBVDNA+] or [HCVRNA+]); Patients with HIV infection or syphilis infection;
6. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systemic AL amyloidosis patients with evaluable hematologic parameter
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Complete hematologic response | 6 months

SECONDARY OUTCOMES:
Overall hematologic response | 6 months
At least one organ response | 12 months
Minimal residual disease | 6 months, 12 months
  Bone marrow miminal residual disease
TTNT | 12 months
  Time to next treatment
MOD-EFS | 12 months
  Major Organ Deterioration Event-Free Survival (MOD-EFS) is defined as the time from the beginning of treatment to hematologic progression, clinical manifestation of end-stage cardiac or renal disease, initiation of subsequent other anti-plasma cell therapy, or death, whichever occur first
MOD-PFS | 12 months
  Major organ deterioration progression-free survival (MOD-PFS) is defined as the time from the beginning of treatment to death, clinical manifestation of end-stage cardiac or renal failure, or hematologic progression, whichever occur first

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Fuxing Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No